CLINICAL TRIAL: NCT03636815
Title: The Effect of Physical Therapy Intervention in Patients With Left Ventricular Assistive Device (LVAD) on Physical Function
Brief Title: The Effect of Physical Therapy Intervention in Patients With Left Ventricular Assistive Device on Physical Function
Acronym: LVAD
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201803106RIND
Record Dates: First submitted 2018-08-01; First posted 2018-08-17 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Left Ventricular Assist Device; Physical Therapy
Keywords: Left ventricular assist device; Physical therapy
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: physical therapy — Cardiopulmonary rehabilitation for patients who receive left ventricle assist device

SUMMARY:
To retrospectively investigate the effect of physical therapy intervention on improving physical function of patients post left ventricular assist device (LVAD) through electronic medical record survey

DETAILED DESCRIPTION:
Method: Using portable electronic medical record system in National Taiwan University Hospital (NTUH), retrospectively survey medical record of patients who underwent left ventricular assist device (LVAD) operation in NTUH, compare improvement among those who had received physical therapy intervention and those who hadn't.

Inclusion criteria: aged older than 20 years old; diagnosed with heart failure and need LVAD implantation

Progress: Note down patients' clinical signs and symptoms, drug usage, imaging findings, physical therapy intervention details, and recovery of functional status. Physical therapy intervention details include: onset symptoms, history, treatment frequency, treatment type, any signs and symptoms during treatment progress and recovery of functional status post physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with heart failure, need left ventricular assist device intervention
* Over 20 years old
* Received physical therapy intervention

Exclusion Criteria:

* N/A

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are diagnosed with heart failure, need left ventricular assist device intervention, and received physical therapy intervention
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2018-04-08 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
Change in walking function | Baseline, two weeks
  By using Six-Minute Walk Test (6MWT), we can obtain the maximum distance that patient can afford walking. In 6 minutes, they should walk as many as they can, on a 15-meter level corridor, assisted device (e.g. cane) can be used if they need. During the test, the patient can stop or rest if they want.

SECONDARY OUTCOMES:
Change in Rating Perceived Exertion (RPE) | Baseline, two weeks
  By using the Borg Rating of Perceived Exertion Scale (score 6-20), the patient subjectively grade the level of perceived exertion after 6MWT.
Change in heart rate | Baseline, two weeks
  While doing 6MWT, patients' heart rate will be monitored through portable electrocardiography (ECG) throughout the test. Resting heart rate and heart rate after 6MWT will be recorded.
Change in blood pressure | Baseline, two weeks
  Resting blood pressure and blood pressure after 6MWT will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University, College of Medicine, Department of Physical Therapy, Taipei, Zhongzheng, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hayes K, Leet AS, Bradley SJ, Holland AE. Effects of exercise training on exercise capacity and quality of life in patients with a left ventricular assist device: a preliminary randomized controlled trial. J Heart Lung Transplant. 2012 Jul;31(7):729-34. doi: 10.1016/j.healun.2012.02.021. Epub 2012 Mar 14. PMID 22425235
- [Background] Kerrigan DJ, Williams CT, Ehrman JK, Saval MA, Bronsteen K, Schairer JR, Swaffer M, Brawner CA, Lanfear DE, Selektor Y, Velez M, Tita C, Keteyian SJ. Cardiac rehabilitation improves functional capacity and patient-reported health status in patients with continuous-flow left ventricular assist devices: the Rehab-VAD randomized controlled trial. JACC Heart Fail. 2014 Dec;2(6):653-9. doi: 10.1016/j.jchf.2014.06.011. Epub 2014 Oct 22. PMID 25447348
- [Background] Laoutaris ID, Dritsas A, Adamopoulos S, Manginas A, Gouziouta A, Kallistratos MS, Koulopoulou M, Voudris V, Cokkinos DV, Sfirakis P. Benefits of physical training on exercise capacity, inspiratory muscle function, and quality of life in patients with ventricular assist devices long-term postimplantation. Eur J Cardiovasc Prev Rehabil. 2011 Feb;18(1):33-40. doi: 10.1097/HJR.0b013e32833c0320. PMID 20571404